CLINICAL TRIAL: NCT05429346
Title: Comparative Effectiveness of Treating Genital Herpes Infection to Reduce Racial Disparities in the Risk of Severe Maternal Morbidity (SMM)
Brief Title: Treating Genital Herpes Infection to Reduce Racial Disparities in the Risk of Severe Maternal Morbidity
Acronym: PCORISMM
Status: Recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1873689
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Genital Herpes Simplex; Maternal Morbidity; Racial Disparities
Keywords: GHSV; SMM; Racial Disparities
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Genital herpes treated before third trimester: Pregnant women with genital herpes infection receiving treatment before the 3rd trimester.
- Genital herpes treated during third trimester: Pregnant women with genital herpes infection receiving treatment during the 3rd trimester.
- Genital herpes untreated: Pregnant women with untreated genital herpes infection.
- Control Group: Pregnant women (controls) with neither genital herpes infection nor treatment.

SUMMARY:
Severe Maternal Morbidity (SMM) has been associated with maternal mortality, fetal risk, and long-term maternal risk. African American (AA) women are at consistently higher risk than White women. However, factors contributing to these racial disparities are largely unknown and commonly known factors have not been able to explain them, so strategies to reduce them are absent. CDC reports that the rate of GHSV infection is 4 times higher in AA than White women. Studies have shown that pregnant women with genital herpes simplex virus (GHSV) infection are at higher risk of SMM and that treating women with GHSV using existing anti-herpes medications could reduce SMM risk. To address the question of racial disparities in SMM and examine the comparative effectiveness of treating women with GHSV infection to reduce the risk of SMM, the investigators are conducting a large cohort study with a two-stage design, combining an EMR-based cohort (Stage I) with a sub-cohort interview (Stage II) to examine the impact of confounders not available from EMR data. Based on status of GHSV and treatment, 4 cohorts of women will be established: (1) those with GHSV infection receiving treatment early in pregnancy; (2) those with GHSV infection receiving treatment later in pregnancy; (3) those with GHSV infection untreated during pregnancy; and (4) those without GHSV. Given that racial disparities in SMM present serious challenges, the study will provide much needed data to address the effectiveness of treating GHSV on reducing racial disparities in SMM.

DETAILED DESCRIPTION:
Severe Maternal Morbidity (SMM), as defined by the CDC, has been repeatedly associated with maternal mortality, fetal risk, and long-term maternal risk. SMM is one of PCORI's research priorities (Special Areas of Emphasis, SAE). Racial disparities in SMM have also been well established, with African American (AA) women having more than twice the risk of SMM than White women However, factors contributing to racial disparities in SMM are largely unknown. Commonly known socio-economic factors have not been able to explain these racial disparities. Due to a lack of understanding of factors contributing to racial disparities in SMM, strategies to reduce them are largely absent.

Recent studies have shown that pregnant women with genital herpes simplex virus (GHSV) infection are at higher risk of pregnancy complications, including SMM. This reported association is supported by strong biological plausibility. Once infected, the virus remains in the body permanently, shedding the virus periodically and causing inflammation in the reproductive tract. The virus is often reactivated during pregnancy due to stress, hormonal changes, and weakened immunity, exacerbating existing inflammation and leading to pregnancy complications, including SMM. At the same time, CDC reports have repeatedly shown that the rate of GHSV infection is 4 times higher in AA women than in White women. Thus, the combination of (a) an increased risk of SMM associated with GHSV infection with (b) high GHSV infection rate in AA makes GHSV a likely contributing factor to the persistently observed racial disparities in SMM. More importantly, recent studies, including a pilot study conducted by the investigators, have shown that treating women with GHSV infection using existing anti-herpes medications could lead to reduction in the risk of SMM. Given that it would benefit AA women more because of their higher GHSV infection rate, the treatment could consequently lead to reduction in racial disparities in SMM. Currently, there is a significant knowledge gap regarding the benefit of treating GHSV infection to reduce the risk of SMM and its racial disparities. Thus, pregnant women with GHSV infection, including many AA women, are not being treated during pregnancy. The current CDC guidelines for treating GHSV infection at 36 weeks of gestation are focused on reducing vertical transmission to newborns; thus, the treatment timing is too late to prevent SMM. Thus, a potentially effective treatment in reducing racial disparities in SMM is not being implemented because of the lack of evidence and the knowledge gap which urgently need to be addressed.

To investigate the comparative effectiveness of treating women with GHSV infection, in comparison to not treating or treating too late, to reduce racial disparities in SMM, the investigators will conduct a large cohort study by leveraging their experience and expertise in studying GHSV infection during pregnancy. The study will consist of pregnant women in four cohorts: (1) women with GHSV infection who received treatment early in pregnancy (before the 3rd trimester); (2) women with GHSV infection who received treatment later in pregnancy (during the 3rd trimester); (3) women with GHSV infection without treatment during pregnancy (untreated); and (4) women without GHSV infection (unexposed controls). Data on GHSV infection and its treatment, SMM diagnosis, and potential confounders are available for all included women from electronic medical records (EMRs). In addition, the study will consist of a sub-cohort of 1,200 participants, selected from each of the four cohorts, who will be interviewed to collect data on additional confounders not available from the EMR. These data will allow the investigators to assess the existence of unmeasured confounders and whether they will impact the results, if any.

The specific aims will address these questions:

Aim 1: Is treating GHSV infection in pregnancy effective in mitigating the racial disparities in SMM? Aim 2: Is treating GHSV infection early in pregnancy more effective than later in pregnancy to mitigate the racial disparities in SMM? Aim 3: Does GHSV infection, if untreated, contribute to racial disparities in the risk of SMM?

The proposed study will address not only one of PCORI research priorities (SAE) in relation to severe maternal morbidity, but also another PCORI priority: reducing racial disparities in health outcomes. The study is also rooted in, and supported by, promising preliminary results and emerging literature with biological plausibility (scientific premise). Unlikely other factors that may contribute to racial disparities that are either very difficult to modify (e.g. sociodemographic factors) or impossible to modify (e.g., genetic factors), if the findings of the pilot study are confirmed, GHSV infection is a modifiable factor that can be treated by existing anti-herpes medications. Thus, the study will fill a knowledge gap which could lead to reduction in racial disparities in SMM through changes in clinical practice of how GHSV infection is treated among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Northern California Members
* Pregnant women

Exclusion Criteria:

* Non Kaiser Permanente Northern California Members
* Non-pregnant women

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All KPNC pregnant women during the study period will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 339000 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Women with SMM | During labor and delivery
  SMM Diagnoses based on CDC's list of 21 indicators

CONTACTS AND LOCATIONS:
Overall Officials: De-Kun Li, MD, PhD, Principal Investigator — Division of Research, Kaiser Permanente Northern California
Locations (1):
- Division of Research, Kaiser Permanente Northern California, Oakland, California, United States